CLINICAL TRIAL: NCT02693470
Title: The Difference of Circulating Endothelial-derived and Platelet-derived Microparticles in Patients With Psoriasis Successfully Treated With Stelara(Ustekinumab)
Brief Title: The Difference of Microparticles in Patients With Psoriasis Vulgaris Who Received Stelara(Ustekinumab)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGMH-0312A3
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Psoriasis With Cell-derived Microparticles
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single-arm study (Other): 50 patients with severe psoriasis who received Stelara(ustekinumab) at 0 and 1 month. The investigators check microparticles level at baseline and 4 months later.
  50 patients without psoriasis: the microparticles are checked at baseline.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — 50 patients with severe psoriasis received ustekinumab 45mg at 0 and 1 month. There were 50 healthy controls. The levels of circulating CD31 and CD41a positive microparticles are measured. In patients with psoriasis, the investigators measure microparticles in the baseline and 4 months after ustekinumab. For control group, the investigators measure microparticles in the baseline.
  Other Names: Stelara

SUMMARY:
Background: Psoriasis, a common inflammatory disease, is associated with atherosclerotic vascular diseases, including stroke, myocardial infarction, and impaired microcirculations, among which circulating microparticles play an important role. In severe psoriasis, there are increased endothelial- and platelet- microparticles that are reduced by TNF-α blockers in parallel with clinical improvement. However, whether Stelara(ustekinumab) treatment would decrease the level of microparticles remains unknown.

Objective: The investigators will evaluate the level of microparticles among normal control, severe psoriasis before and 4 months after ustekinumab treatment.

DETAILED DESCRIPTION:
Methods: The investigators will recruit 50 patients with severe psoriasis who received ustekinumab and 50 control subjects without psoriasis from August 2014 to July 2016. Concentrations of microparticles with expression for surface markers (Annexin V, CD31, and CD41a) will be measured in peripheral blood using flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe psoriasis who receive ustekinumab treatment.
* Patients in the control group are examined thoroughly to make sure no psoriatic lesions by two dermatologists. Age, sex, lipid profiles, and blood pressure are recorded for all subjects.

Exclusion Criteria:

* The psoriatic patients and healthy controls who have pregnancy or infection (such as tuberculosis or sepsis) are excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
The difference of CD41a and CD31 positive microparticles in patients with severe psoriasis before and after ustekinumab treatment. | The levels of CD41a and CD31 positive microparticles are checked in patients with psoriasis before and 4 months after ustekinumab.

SECONDARY OUTCOMES:
The difference of CD41a and CD31 positive microparticles between normal control and patients with severe psoriasis | Patients with severe psoriasis: microparticles are checked at baseline. Control group: microparticles are checked at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Lee, M.D.PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Department of Dermatology, Kaohsiung Chang Gung Memorial Hospital and Chang Gung University College of Medicine, Kaohsiung, Taiwan, Kaohsiung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No